CLINICAL TRIAL: NCT03858764
Title: Local Paclitaxel Delivery to Prevent Restenosis Using the TAPAS Catheter After Endovascular Revascularization in Patients With Previous Femoropopliteal Intervention
Brief Title: Local Paclitaxel Delivery to Prevent Restenosis in Peripheral Arterial Disease
Acronym: ResTAP
Status: Withdrawn | Type: Observational
Why Stopped: no patients enrolled. primary investigator never started study
Sponsor: Jane Phillips Medical Center (Other)
Responsible Party: Principal Investigator, Anderson Mehrle M.D., Interventional Cardiologist, Jane Phillips Medical Center
Other Study IDs: APMABR 7181
Record Dates: First submitted 2018-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Arterial Disease; Restenosis
Keywords: Paclitaxel; Peripheral arterial disease; restenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

SUMMARY:
The purpose of this study is to determine if the addition of a catheter-based local delivery of paclitaxel into the peripheral arterial vessels in patients with peripheral arterial disease (PAD) and subsequent restenosis of the femoropopliteal region would benefit from this type of investigational intervention with a known antiproliferative agent.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) of the lower extremities is an extremely prevalent, and often times, disabling disorder reaching roughly 8 million people in the United States, and up to 20 percent of the population over the age of 60 to 70. Atherosclerosis commonly occurs in the superficial femoral artery (SFA) and the popliteal artery limiting blood flow to the affected vessels, as well as, the distal lower extremities. PAD of this type causes claudication in up to 35% of patients which may progress to critical limb ischemia in up to 2%.

Endovascular treatment options have significantly improved over the past decade, allowing a multitude of treatment alternatives. In the US, the number of endovascular treatments now exceed bypass surgery. Procedural success rates of greater than 90 percent can be achieved by stenting, atherectomy, and percutaneous transluminal angioplasty; however, long term patency rates have been troubled by elastic recoil or neointimal hyperplasia. Two year patency rates have been documented to range from 40-50% following balloon angioplasty. Stenting in the femoropopliteal region in attempts to improve restenosis fall short with a primary patency rate of 70-80% as seen in the FAST trial. Atherectomy is promising, but has not been studied extensively.

The inability to obtain long term patency has led us to look at our success in the coronary field where drug-eluting stents (DES) are often used. Antiproliferative drugs such as paclitaxel prevent neointimal growth and have proven patency and long term success. There have been initial animal and human studies which have shown potential in preventing restenosis by using drug coated balloons and DES. Currently, there is no FDA approved drug eluting balloon for use in femoropopliteal disease, leading us to search for alternative therapies following femoropopliteal interventions.

Paclitaxel inhibits microtubule disassembly and disrupts normal cellular processes such as protein signaling, mitosis, and migration. It is highly lipogenic and poorly water soluble. Paclitaxel has been stated to prevent restenosis through several mechanisms in vitro. These mechanisms include inhibiting proliferation and migration of human smooth muscle cells. Use of the antiproliferative agent in the peripheral arena has been conducted, but no definitive results have been achieved to date. One internal animal study showed promise in the deliverability of localized paclitaxel into targeted segments of the vessel using the TAPAS device. Concentrations of 0.67 mg/mL, 1.2 mg/mL, and 2.0 mg/mL were infused locally at a duration of 2-5 minutes within the iliofemoral segment in pigs, then aspirated from the vessel using the device. No differences in drug absorption were found among the three concentrations. Drug retention remained greater than 50% in all groups at 3 and 24 hours. The average drug concentration in the vessel wall of all groups was 1.73 ± 0.85 µg/g at 3 hours, and 1.29 ± 0.47 µg/g at 24 hours after treatment. Approximately 77% of the total drug administered was aspirated, with the assumption that the remaining drug was either absorbed in the tissue, remained in the catheter, or lost systemically. On average, plasma paclitaxel levels after treatment measured 22.5 ± 21.07 ng/mL at 2 minutes, 2.7 ± 0.85 ng/mL at 3 hours, and less than 1.2 ng/mL at 24 hours. Histology showed no inflammation, injury, or other adverse effect when compared with the contrast group.

The newly available Targeted Adjustable Pharmaceutical Application System (TAPAS)-TAPAS Catheter Therapeutic System (Spectranetics, Colorado Springs, CO, USA)-has a proximal and distal occlusion balloon with an adjustable length that allows local drug delivery to a targeted arterial segment preventing systemic effects by allowing aspiration following delivery.

The ResTAP study is a prospective, open label, observational study to assess the safety and efficacy of the delivery of paclitaxel to prevent recurrent restenosis after percutaneous intervention including atherectomy with or without stenting in patients who have restenosis after a prior endovascular revascularization.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Rutherford Stages 2-5 plus prior history of endovascular revascularization and recurrent stenosis (in stent, post angioplasty, post atherectomy) (Table 1 )
* one or more restenotic lesions within the SFA of at least 70% of the vessel diameter
* Successful percutaneous revascularization of the femoropopliteal artery (< 20% residual stenosis by visual estimate) using standard techniques per discretion of the local operator
* The femoropopliteal Reference Vessel Diameter (RVD) must be ≥4.0 mm and ≤7.0 mm

Exclusion Criteria:

* Patient is pregnant or breast feeding. (Female subjects of childbearing potential must have negative serum pregnancy test the day of the procedure.)
* Life expectancy < 12 months.
* Contraindication to aspirin, clopidogrel or other thienopyridine, heparin, low molecular weight heparin, bivalirudin or other therapies required for procedure or follow up.
* Known allergy to contrast media that cannot adequately be pre-medicated prior to study procedure.
* Known allergy to paclitaxel.
* Uncontrolled hypercoagulability or history of HIT or HITTS syndrome.
* Simultaneous enrollment in another investigational device or drug study.
* Absence of at least 1 TIMI-3 vessel run off into the foot.
* Platelet count < 100,000/mm3.
* White blood cell count < 1.5/mm3.
* Any evidence of perforation or dye extravasation during the index procedure, even if successfully treated with a covered stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with peripheral arterial disease and subsequent restenosis of the previously treated femoropopliteal region seen in either the Bluestem Cardiology Office or at Jane Phillips Medical Center under the care of one of the Bluestem cardiologists
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Primary Patency | 6 months
  Loss of primary patency will occur for any clinically driven Target Lesion Revascularization (TLR) as determined by Rutherford scale on claudication and a Peak Systolic Velocity Ratio (PSVR) of > 2.5 on Duplex Ultrasound (DUS), or CTA quantified stenosis ≥ 70%
Primary Safety | 1 month
  Freedom from death, major amputation in the target limb, or Target Lesion Revascularization (either surgical or endovascular)

SECONDARY OUTCOMES:
Primary Patency | 1, 3, and 12 months
  Loss of primary patency will occur for any clinically driven Target Lesion Revascularization (TLR) or a Peak Systolic Velocity Ratio (PSVR) of > 2.5 on Duplex Ultrasound (DUS), CTA quantified stenosis ≥ 70%
Primary Assisted Patency | 6, 12 months
  Patency of the target vessel regardless of secondary interventions performed to restore blood flow after restenosis.
Secondary Patency | 6, 12 months
  Patency of the target vessel regardless of secondary interventions performed to restore blood flow after re-occlusion
Functional Status | 1, 3, 6, and 12 months
  Rutherford Classification
Secondary Safety | 1, 3, 6, 12 months
  adverse events associated with the use of paclitaxel, such as, but not limited to: hypotension, anaphylactic reactions, nausea, vomiting, diarrhea pancytopenia, neuropathy, alopecia which will be determined by clinical assessment and review of systems at time of exam